CLINICAL TRIAL: NCT03214757
Title: A Study of Impact of Anemia on Morbidity and Mortality in Children With Dilated Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Amar, principal investigator, Assiut University
Other Study IDs: NA_0000XXX
Record Dates: First submitted 2017-07-07; First posted 2017-07-12 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Pediatric Dilated Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group with dilated cardiomyopathy without anemia
- group with dilated cardiomyopathy with anemia
  Interventions: Other: treatment of anemia.

INTERVENTIONS:
Other: treatment of anemia. — drug treatment of anemia.
  Groups: group with dilated cardiomyopathy with anemia

SUMMARY:
Dilated cardiomyopathy is a heart muscle disorder characterized by systolic dysfunction and dilation of the left or both ventricles.Dilated cardiomyopathy can develop in people of any age or ethnicity, although it is more common in male than female persons occurring at a ratio of about three to one in male to female persons.

Dilated cardiomyopathy is the predominant cause of cardiomyopathy in pediatric populations. Annual incidence in pediatric populations has been reported to be much lower than one to one hundred seventy thousand in the United States and one to one hundred forty thousand in Australia.

Although pediatric dilated cardiomyopathy has a lower annual incidence than adult dilated cardiomyopathy, the outcome for pediatric dilated cardiomyopathy patients is particularly severe.

Dilated cardiomyopathy is the most frequent cause of heart transplantation in pediatric patients. Data from international pediatric dilated cardiomyopathy registries indicate that the rates of death or heart transplantation over one and five year periods were thirty one percent and forty six percent, respectively.

Onset of dilated cardiomyopathy is usually insidious but may be acute in as many at twenty five percent of patients. Approximately fifty percent of patients with dilated cardiomyopathy have a history of preceding viral illness.

DETAILED DESCRIPTION:
The clinical diagnosis of dilated cardiomyopathy is made from history, physical examination, and noninvasive testing. The initial clinical manifestations of dilated heart failure are generally those of respiratory distress secondary to congestion of the pulmonary and systemic venous circulations.

Pallor, irritability, diaphoresis, tachypnea, easy fatigability are characteristics.

Failure to grow may also occur. In older patients, a history of orthopnea, nocturnal cough, and dyspnea provoked by minimal activity can be elicited and generally precede evidence of systemic venous congestion. In rapidly progressive disease, dominant symptoms are often abdominal distention, right upper quadrant pain, and nausea. Less often, initial symptoms in childhood include arrhythmias, syncope, neurologic problems (seizures or delayed development), vomiting, abdominal distention, or fever.

Although as many as fifty percent of children with cardiomyopathy and heart failure give a history of a nonspecific febrile illness within three months of presentation, no evidence of myocarditis can usually be found on biopsy.'Physical signs vary with the stage of the disease.

Signs of congestive heart failure are frequent, and include tachypnea,tachycardia, diaphoresis, hepatomegaly, pallor, and, in advanced cases, hypotension and shock.

Failure to thrive may be present if, heart failure has been long standing. Patients are generally not cyanotic. Wheezing may be heard; however, rales are infrequent, especially in infants.

Neck vein distension is common, the external jugular crest reflecting mean right atrial pressure, the internal jugular exhibiting a prominent V wave indicative of tricuspid regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* All infants and children with dilated cardiomyopathy who are diagnosed clinically and by echocardiography attending cardiology outpatient clinic at Assiut University Children Hospital will be included.

Exclusion Criteria:

* Infants age less than two months.
* Infants with hemolytic anemias.
* Patients with congestive heart failure due to congenital heart disease.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All infants and children with dilated cardiomyopathy who are diagnosed clinically and by echocardiography attending cardiology outpatient clinic at Assiut University Children Hospital.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Heart failure | four months duration after start of the study
  Through clinical manifestations of heart of heart failure and echocardiographic assesment of ventricular function

OTHER OUTCOMES:
Quality of Well-Being Scale | three months duration after start of the study
  To measure health related quality of life, to monitor the health of populations over time, or to evaluate the efficacy and effectiveness of clinical therapies of practices using a preference weighted self administered measure.